CLINICAL TRIAL: NCT05292677
Title: Prospective, Single-Blind Randomized Trial of in Office Superior Laryngeal Nerve Block for the Treatment of Chronic Neurogenic Cough
Brief Title: Laryngeal Nerve Block for Chronic Cough
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Benjamin J Rubinstein, Assistant Professor, Eastern Virginia Medical School
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14Jul2021
Record Dates: First submitted 2021-09-14; First posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Laryngeal Nerve Block; Chronic Neurogenic Cough; Laryngeal Hypersensitivity
Keywords: cough; chronic cough; neurogenic cough; laryngeal nerve block
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Steroid/Anesthetic Mixture) (Experimental): The steroid/anesthetic mixture will be injected via a 27-gauge needle once at the baseline or during the 6-week crossover timepoint.
  Interventions: Drug: Steroid/Anesthesia Mixture
- Placebo (Normal Saline) (Placebo Comparator): The placebo (Normal Saline) will be injected via a 27-gauge needle once at the baseline or during the 6-week crossover timepoint.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Steroid/Anesthesia Mixture — Steroid will be Triamcinolone Acetonide (40mg/mL). Anesthetic will be 0.5% bupivacaine with 1:100,000 epinephrine. These will be pre-mixed by a qualified personnel within the ENT department.
  Arms: Intervention (Steroid/Anesthetic Mixture)
Drug: Placebo — 2 mL of Normal Saline
  Arms: Placebo (Normal Saline)

SUMMARY:
The purpose of this study is to study the potential benefit of treating chronic neurogenic cough by blocking the nerve responsible for the disease with an injection of local anesthetic/steroid mixture versus a placebo.

DETAILED DESCRIPTION:
This study will be performed by asking participants to fill out multiple questionnaires on the symptoms of their cough, and undergo cough testing by inhaling an airway irritant and monitoring the number of coughs after inhalation of the irritant. Subjects would then undergo the treatment and have an injection of either local anesthetic/steroid mixture or a placebo (normal saline) around the nerve that gives feeling to the portion of the voice box responsible for chronic neurogenic cough. After the injection you will be asked to repeat the cough testing and questionnaires 30 minutes, 1 weeks, and at 6 weeks post injection. After the initial six weeks, patients will cross over and repeat the same process with the opposite treatment (either local anesthetic/steroid mixture or placebo) from their previous injection. The total time of participation is about 12 weeks and we hope to recruit 40 subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Previously or Newly Diagnosed Chronic Neurogenic Cough

Exclusion Criteria:

* History of Laryngeal Surgery or External Beam Radiation
* Current Smokers
* Known Allergy or Sensitivity to Local Anesthetics
* Uncontrolled Pulmonary, SinoNasal, or GastroIntestinal Pathology leading to Refractory Chronic Cough

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
Intervention vs. Placebo in Neurogenic Cough using Capsaicin Challenge | Comparing Changes at Pretreatment, at 30 minutes post treatment, at 1 week post treatment, and at 6 weeks post treatment
  Objectively evaluate the efficacy of blockade of the internal branch of the superior laryngeal nerve with local anesthetic/steroid mixture compared to normal saline placebo in treating chronic neurogenic cough using capsaicin challenge testing to measure cough sensitivity and urge to cough

SECONDARY OUTCOMES:
Intervention vs. Placebo in Neurogenic Cough using the Newcastle Laryngeal Hypersensitivity Questionnaire | Pretreatment, 30 minutes post treatment, 1 week post treatment, 6 weeks post treatment
  Subjectively evaluate the efficacy of superior laryngeal nerve block (intervention) vs. placebo using the Newcastle Laryngeal Hypersensitivity Questionnaire (NLHQ). This Questionnaire is scaled from 1 to 7. 1 indicates All of the Time while 7 reflects None of the Time.
Intervention vs. Placebo in Neurogenic Cough using the Urge to Cough Scale | Pretreatment, 30 minutes post treatment, 1 week post treatment, 6 weeks post treatment
  Subjectively evaluate the efficacy of superior laryngeal nerve block (intervention) vs. placebo using the Urge to Cough Scale. Higher score indicates more urge, while lower score reflects less of an urge to cough.
Intervention vs. Placebo in Neurogenic Cough using the Central Sensitization Inventory | Pretreatment, 30 minutes post treatment, 1 week post treatment, 6 weeks post treatment
  Subjectively evaluate the efficacy of superior laryngeal nerve block (intervention) vs. placebo using the Central Sensitization Inventory (CSI). Scale is ranked as Never, Rarely, Sometimes, Often, and Always and has various symptoms listed.
Quality of Life Measurements | Pretreatment, 1 week post treatment, 6 weeks post treatment
  Analyze quality of life measurements of patients undergoing superior laryngeal nerve block compared to placebo as measured by the Leicester Cough Questionnaire (LCQ). Scale is from a 1 to 7. The higher the score/rating represents less of a problem while a lower score/rating represents more of a problem.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Rubinstein, MD, Principal Investigator — Eastern Virginia Medical School Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- Eastern Virginia Medical School Ear, Nose, and Throat Surgeons, Norfolk, Virginia, United States